CLINICAL TRIAL: NCT05768243
Title: Efficiency of Hyaluronic Acid Versus Red Injectable Platelet-Rich Fibrin (i-PRF) in Treatment of Stage III Periodontitis (Randomized Controlled Clinical Trial)
Brief Title: Hyaluronic Acid Versus Red Injectable Platelet Rich Fibrin in Treatment of Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beirut Arab University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-H-0075-D-R-0293
Record Dates: First submitted 2023-02-20; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Periodontitis Chronic Generalized Severe
MeSH Terms: interventions — Hyaluronic Acid; proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treated with hyaluronic acid + SRP (Experimental): After scaling and root planing, hyaluronic acid (GENGIGEL®) will be applied in the following forms (one ml of 0.8% HA was injected subgingivally once every four weeks), topically (0.2 ml of 0.8% HA applied by the patient twice daily for the following 14 days after the subgingival application).
  Interventions: Drug: Hyaluronic acid
- Treated with red i-PRF + SRP (Experimental): The red i-PRF will be injected into the pocket at the point of interdental space after SRP. Moreover, to control bleeding due to the needle tip after the procedure, a saline-soaked sponge will be placed between the lip and the gingiva and removed after 15 minutes. A total of four sessions of i-PRF will be administered to patients at a ten-day interval.
  Interventions: Procedure: red injectable platelet rich fibrin (i-prf)
- Scaling and root planing only (No Intervention): no adjunctive treatment will be done to scaling and root planing

INTERVENTIONS:
Drug: Hyaluronic acid — hyaluronic acid is used as an adjunctive treatment to scaling and root planing
  Other Names: GENGIGEL®
  Arms: Treated with hyaluronic acid + SRP
Procedure: red injectable platelet rich fibrin (i-prf) — injecting red i-prf into the pocket after scaling and root planing
  Arms: Treated with red i-PRF + SRP

SUMMARY:
the aim of this clinical trial is to compare the efficacy of hyaluronic acid (HA) used as an adjunctive to scaling and root planing (SRP) and red injectable platelet rich-fibrin (i-PRF) in the non-surgical treatment of stage III periodontitis. The main question it aims to answer is: is there a difference between HA and red i-prf when used as an adjunct to SRP in terms of efficacy?

Participants who are eligible will be assigned to one of the treatment groups:

* Group 1= receives HA+ SRP
* Group 2= receives red i-prf + SRP
* Group 3= receives only SRP

Researchers will compare Groups 1,2 and 3 to see if there's a difference in the periodontal parameters measured.

DETAILED DESCRIPTION:
Complete medical and dental histories as well as informed consent will be collected from eligible participants, and periodontal charting will be done for them.

The selected patients will be allocated into three groups (each containing 25) with the help of a computerized randomizer (Randomizer.org):

* Group one (G1): 25 patients will be treated with hyaluronic acid gel as an adjunct to scaling and root planing by applying one ml of 0.8% HA to the base of the pocket (subgingivally) and 0.2 ml of 0.2% HA topically (applied by the patient).
* Group two (G2): 25 patients will be treated with red i-PRF as an adjunct to scaling and root planing.
* Group three (G3): 25 patients will be treated with scaling and root planing only.

The clinical examiner will not be informed of the treatment groups' distribution.

Before the baseline examination, a full mouth supragingival scaling and root planing will be performed under local anesthesia in one or two sessions (over a 24-hour period). Patients will be informed on self-performed plaque control measures, including using the modified Bass brushing technique using a soft toothbrush and regular toothpaste twice a day and interdental cleaning using interdental brushes once a day. Patients will receive the same toothbrushes, toothpaste, and interdental brushes.

The clinical parameters will be recorded at the baseline (1st visit) before the treatment and will be repeated in the fourth week (2nd visit), eighth week (3rd visit), and twelfth week (fourth visit). During this period, reinforcement of plaque control will be given to maintain good oral hygiene.

Data from previous studies will be used to calculate the sample size (Zijnge et al., 2010) regarding the PD change measurement. It is found that the difference in PD (δ) is around 0.3mm, whereas the standard deviation in groups (σ) is around 0.2mm. Our aim is to achieve a statistical power of > 90% as well as a 0.05 significance level. Thus, 18 participants per group will be needed. However, as some dropouts may be expected, a minimum of 25 patients per group will be recruited.

Statistical analysis will be done using SAS 9.4 Software (SAS Institute Inc., Cary, NC, USA). Means and standard deviations (SD) will be calculated for all continuous variables (periodontal parameters: CAL, PD, BOP, GI, PI) at the baseline, fourth week, eighth week, and twelfth week. Repeated linear mixed-effects models (PROC MIXED in SAS) will be used to examine the changes in all periodontal parameters over the four-time points within each group and between groups. An unstructured covariance matrix will be used, residual plots will be visually reviewed to check model fit, and extreme outliers will be eliminated using the restricted likelihood distance. A Tukey-Kramer correction will be applied to all pairwise comparisons. One-way ANOVA is to be used to examine group differences in PD reduction and CAL. A p-value of 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* clinical periodontal loss and radiographic bone loss of stage III/grades A and B with no history of systemic disease.
* at least four periodontal sites with a pocket depth of six mm or greater
* radiographic evidence of bone loss extending to the middle third of the root
* clinical attachment loss of five mm or more

Exclusion Criteria:

* uncontrolled systemic conditions (uncontrolled diabetes or uncontrolled hypertension)
* bleeding disorders, or on anticoagulant therapy
* alcohol users
* pregnant or lactating females
* heavy smokers (more than ten cigarettes per day)
* chemo or radio therapy
* antibiotic/anti-inflammatory drugs over the last three months before treatment.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-24 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level | 4 weeks
  used to assess the loss of periodontal tissue support in periodontitis. It is the distance from the cemento-enamel junction (fixed point on the tooth) to the depth of the pocket
Probing Depth | 4 weeks
  used to detect the depth of the periodontal pocket. It is the distance from the gingival margin to the base of the pocket.

SECONDARY OUTCOMES:
Bleeding on Probing | 4 weeks
  It is an indicator of periodontal tissue inflammatory response. The probe is carefully introduced to the bottom of the pocket and gently moved laterally along the pocket wall. Depending on the severity of inflammation, bleeding can vary from a tenuous red line along the gingival sulcus to profuse bleeding (immediately after probing or few seconds after).
Plaque index | 4 weeks
  used to evaluate the level and rate of plaque formation on tooth surfaces. It measures the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth, except the third molars. The amount of plaque is determined with disclosing solution and a range of scores of 0-5 is assigned with 0 denoting no plaque and 5 denoting heavy plaque (covering 2/3 of the tooth crown)
Gingival index | 4 weeks
  used to assess the severity of gingival inflammation. Scores ranges from 0-3 with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling, and spontaneous bleeding. This measurement is based on the presence or absence of bleeding on gentle probing

CONTACTS AND LOCATIONS:
Overall Officials: Nayer Aboelsaad, PhD, Study Chair — Professor and Chairman of Periodontology department - BeirutArabU
Locations (1):
- Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dietrich T, Ower P, Tank M, West NX, Walter C, Needleman I, Hughes FJ, Wadia R, Milward MR, Hodge PJ, Chapple ILC; British Society of Periodontology. Periodontal diagnosis in the context of the 2017 classification system of periodontal diseases and conditions - implementation in clinical practice. Br Dent J. 2019 Jan 11;226(1):16-22. doi: 10.1038/sj.bdj.2019.3. PMID 30631188
- [Background] Dahiya P, Kamal R. Hyaluronic Acid: a boon in periodontal therapy. N Am J Med Sci. 2013 May;5(5):309-15. doi: 10.4103/1947-2714.112473. PMID 23814761
- [Background] Sanz I, Alonso B, Carasol M, Herrera D, Sanz M. Nonsurgical treatment of periodontitis. J Evid Based Dent Pract. 2012 Sep;12(3 Suppl):76-86. doi: 10.1016/S1532-3382(12)70019-2. PMID 23040340
- [Background] Casale M, Moffa A, Vella P, Sabatino L, Capuano F, Salvinelli B, Lopez MA, Carinci F, Salvinelli F. Hyaluronic acid: Perspectives in dentistry. A systematic review. Int J Immunopathol Pharmacol. 2016 Dec;29(4):572-582. doi: 10.1177/0394632016652906. Epub 2016 Jun 8. PMID 27280412
- [Background] Hakkinen L, Uitto VJ, Larjava H. Cell biology of gingival wound healing. Periodontol 2000. 2000 Oct;24:127-52. No abstract available. PMID 11276865
- [Background] Kour P, Pudakalkatti PS, Vas AM, Das S, Padmanabhan S. Comparative Evaluation of Antimicrobial Efficacy of Platelet-rich Plasma, Platelet-rich Fibrin, and Injectable Platelet-rich Fibrin on the Standard Strains of Porphyromonas gingivalis and Aggregatibacter actinomycetemcomitans. Contemp Clin Dent. 2018 Sep;9(Suppl 2):S325-S330. doi: 10.4103/ccd.ccd_367_18. PMID 30294166
- [Background] Thanasrisuebwong P, Kiattavorncharoen S, Surarit R, Phruksaniyom C, Ruangsawasdi N. Red and Yellow Injectable Platelet-Rich Fibrin Demonstrated Differential Effects on Periodontal Ligament Stem Cell Proliferation, Migration, and Osteogenic Differentiation. Int J Mol Sci. 2020 Jul 21;21(14):5153. doi: 10.3390/ijms21145153. PMID 32708242
- [Background] Xu Y, Hofling K, Fimmers R, Frentzen M, Jervoe-Storm PM. Clinical and microbiological effects of topical subgingival application of hyaluronic acid gel adjunctive to scaling and root planing in the treatment of chronic periodontitis. J Periodontol. 2004 Aug;75(8):1114-8. doi: 10.1902/jop.2004.75.8.1114. PMID 15455740
- [Background] Gontiya G, Galgali SR. Effect of hyaluronan on periodontitis: A clinical and histological study. J Indian Soc Periodontol. 2012 Apr;16(2):184-92. doi: 10.4103/0972-124X.99260. PMID 23055583
- [Background] Aydinyurt HS, Akbal D, Altindal D, Bozoglan A, Ertugrul AS, Demir H. Evaluation of biochemical and clinical effects of hyaluronic acid on non-surgical periodontal treatment: a randomized controlled trial. Ir J Med Sci. 2020 Nov;189(4):1485-1494. doi: 10.1007/s11845-020-02230-6. Epub 2020 May 21. PMID 32436173
- [Background] Vanden Bogaerde L. Treatment of infrabony periodontal defects with esterified hyaluronic acid: clinical report of 19 consecutive lesions. Int J Periodontics Restorative Dent. 2009 Jun;29(3):315-23. PMID 19537471
- [Background] Johannsen A, Tellefsen M, Wikesjo U, Johannsen G. Local delivery of hyaluronan as an adjunct to scaling and root planing in the treatment of chronic periodontitis. J Periodontol. 2009 Sep;80(9):1493-7. doi: 10.1902/jop.2009.090128. PMID 19722800
- [Background] Pilloni A, Annibali S, Dominici F, Di Paolo C, Papa M, Cassini MA, Polimeni A. Evaluation of the efficacy of an hyaluronic acid-based biogel on periodontal clinical parameters. A randomized-controlled clinical pilot study. Ann Stomatol (Roma). 2011 Mar;2(3-4):3-9. Epub 2012 Jan 27. PMID 22545183
- [Background] Karakostas P, Davidopoulou S, Kalfas S. Use of Hyaluronic Acid in Periodontal Disease Treatment: A Systematic Review. J Contemp Dent Pract. 2022 Mar 1;23(3):355-370. PMID 35781443
- [Background] Olszewska-Czyz I, Kralik K, Tota M, Prpic J. The Influence of Hyaluronic Acid Adjunctive Therapy of Periodontitis on Salivary Markers of Oxidative Stress: Randomized, Controlled Clinical Trial. Antioxidants (Basel). 2022 Jan 7;11(1):135. doi: 10.3390/antiox11010135. PMID 35052639
- [Background] Yan Y, Zhan Y, Wang X, Hou J. Clinical evaluation of ultrasonic subgingival debridement versus ultrasonic subgingival scaling combined with manual root planing in the treatment of periodontitis: study protocol for a randomized controlled trial. Trials. 2020 Jan 28;21(1):113. doi: 10.1186/s13063-019-4031-y. PMID 31992331
- [Background] Zijnge V, Meijer HF, Lie MA, Tromp JA, Degener JE, Harmsen HJ, Abbas F. The recolonization hypothesis in a full-mouth or multiple-session treatment protocol: a blinded, randomized clinical trial. J Clin Periodontol. 2010 Jun;37(6):518-25. doi: 10.1111/j.1600-051X.2010.01562.x. PMID 20507375
- [Background] Wang X, Zhang Y, Choukroun J, Ghanaati S, Miron RJ. Behavior of Gingival Fibroblasts on Titanium Implant Surfaces in Combination with either Injectable-PRF or PRP. Int J Mol Sci. 2017 Feb 4;18(2):331. doi: 10.3390/ijms18020331. PMID 28165420
- [Background] Thanasrisuebwong P, Surarit R, Bencharit S, Ruangsawasdi N. Influence of Fractionation Methods on Physical and Biological Properties of Injectable Platelet-Rich Fibrin: An Exploratory Study. Int J Mol Sci. 2019 Apr 3;20(7):1657. doi: 10.3390/ijms20071657. PMID 30987117
- [Background] Fang H, Han M, Li QL, Cao CY, Xia R, Zhang ZH. Comparison of full-mouth disinfection and quadrant-wise scaling in the treatment of adult chronic periodontitis: a systematic review and meta-analysis. J Periodontal Res. 2016 Aug;51(4):417-30. doi: 10.1111/jre.12326. Epub 2015 Oct 19. PMID 26477533
- See also: accepted paper (yet not published in a journal) — http://doi.org/10.2298/SARH190925022V

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT05768243/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT05768243/ICF_001.pdf